CLINICAL TRIAL: NCT03562338
Title: Modelo Preditivo Para os Resultados de Sucesso Com um Programa Combinado de Terapia Manual e exercício em indivíduos Com Dor Cervical crónica de Origem não-especifica
Brief Title: Predictive Model of Recovery in Patients With Chronic Nonspecific Neck Pain Undergoing Manual Therapy and Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: NOVA.MS|FCM-UNL
Record Dates: First submitted 2018-05-24; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Chronic Nonspecific Neck Pain
Keywords: chronic nonspecific neck pain; disability; predictive model; rehabilitation; pain intensity
MeSH Terms: conditions — Pain | interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy and Exercise (Experimental)
  Interventions: Other: Manual Therapy and Exercise (Physiotherapy Intervention)
- Usual Care (Active Comparator)
  Interventions: Other: Usual Care (Physiotherapy Intervention)

INTERVENTIONS:
Other: Manual Therapy and Exercise (Physiotherapy Intervention) — Participants in this group will receive a 6-weeks program of mobilization and progressive exercise for the neck flexors, 2 times a week.
  Arms: Manual Therapy and Exercise
Other: Usual Care (Physiotherapy Intervention) — Participants in this group will receive usual care in physiotherapy during the 6-weeks period.
  Arms: Usual Care

SUMMARY:
The aim of this study is to develop a predictive model to identify which patients with chronic nonspecific neck pain are more likely to benefit from manual therapy and exercise program, or usual care.

ELIGIBILITY:
Inclusion Criteria:

* Chronic nonspecific neck pain at least 3 months, defined as pain in the cervical region without a specific anatomopathological diagnosis;
* Adults between 18 and 65 years of age and literate in Portuguese;

Exclusion Criteria:

* History of cervical trauma and/or history of surgery in the prior 6 months;
* Clinical signs of infection, tumor, neurological, inflammatory or systemic diseases;
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-06-11 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Neck Pain Intensity as measured by the Numeric pain rating scale (NRPS) at 3 weeks. | 3 weeks
  The change will be defined on the Minimal Clinically Important Difference in treatment response defined as a decrease of ≥2 point in NRPS (range: 0 - 10 points).
Change from baseline in Neck Pain Intensity as measured by the Numeric pain rating scale (NRPS) at 6 weeks. | 6 weeks
  The change will be defined on the Minimal Clinically Important Difference in treatment response defined as a decrease of ≥2 point in NRPS (range: 0 - 10 points).
Change from baseline in Neck Pain Intensity as measured by the Numeric pain rating scale (NRPS) at follow-up 3 months. | Follow-up 3 months
  The change will be defined on the Minimal Clinically Important Difference in treatment response defined as a decrease of ≥2 point in NRPS (range: 0 - 10 points).
Change from baseline in Neck Disability as measured by the Neck Disability Index (NDI) at 3 weeks. | 3 weeks
  The change will be defined on the Minimal Clinically Important Difference in treatment response defined as a decrease of ≥27% in NDI (range: 0-50 and higher scores are indicative of more disability).
Change from baseline in Neck Disability as measured by the Neck Disability Index (NDI) at 6 weeks. | 6 weeks
  The change will be defined on the Minimal Clinically Important Difference in treatment response defined as a decrease of ≥27% in NDI (range: 0-50 and higher scores are indicative of more disability).
Change from baseline in Neck Disability as measured by the Neck Disability Index (NDI) at follow-up 3 months. | Follow-up 3 months
  The change will be defined on the Minimal Clinically Important Difference in treatment response defined as a decrease of ≥27% in NDI (range: 0-50 and higher scores are indicative of more disability).

SECONDARY OUTCOMES:
Clinical Important Treatment response in global perceived recovery as measured by Patient's Global Impression of Change Scale at 3 weeks | 3 weeks
  The clinically Important treatment response in global perceived recovery was defined as a value of ≥5 in Patient's Global Impression of Change Scale (range: 1-7 Likert Scale)
Clinical Important Treatment response in global perceived recovery as measured by Patient's Global Impression of Change Scale at 6 weeks | 6 weeks
  The clinically Important treatment response in global perceived recovery was defined as a value of ≥5 in Patient's Global Impression of Change Scale (range: 1-7 Likert Scale)
Clinical Important Treatment response in global perceived recovery as measured by Patient's Global Impression of Change Scale at follow-up 3 months | Follow-up 3 months
  The clinically Important treatment response in global perceived recovery was defined as a value of ≥5 in Patient's Global Impression of Change Scale (range: 1-7 Likert Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Lúcia Domingues, Principal Investigator — NOVA Medical School | Faculdade de Ciências Médicas, Universidade Nova de Lisboa